CLINICAL TRIAL: NCT07256639
Title: Evaluating Heart & Soil's Whole Package on Men's Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 41342
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Testosterone

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single arm where participants act as their own control
  Interventions: Dietary Supplement: Heart and Soil's Whole Package

INTERVENTIONS:
Dietary Supplement: Heart and Soil's Whole Package — Whole Package is a male health supporting supplement made of 100% grass-fed beef liver, testicle, and whole blood extract.

SUMMARY:
This study explores how Heart & Soil's Whole Package impacts men's hormone health, strength, and virility using blood testosterone tracking and self-reported measures.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to meticulously investigate the role of organ-derived supplements, specifically Heart & Soil's Whole Package, in influencing male hormone health, particularly testosterone levels, and aspects of virility including mood, muscle mass, performance, and overall vitality. Despite the widespread use of both natural and synthetic supplements to enhance male health, the scientific community has paid little attention to the potential benefits of organ-derived supplements. Heart & Soil has gathered numerous anecdotal reports from users of Whole Package, who have experienced notable improvements in energy, strength, libido, and general well-being. This research aims to bridge this knowledge gap by applying a rigorous scientific approach to evaluate the effects of Whole Package supplementation on men's hormonal balance and virility.

Participants in this study will undergo a comprehensive evaluation of their health status, focusing on blood testosterone levels and self-reported measures of male virility, both before and after the supplementation period. This approach allows for a personalized analysis of how Whole Package might contribute to male hormone health and performance enhancements. By collecting and analyzing data on changes in testosterone levels and other virility indicators, investigators seek to provide participants with individualized insights into the potential health benefits of incorporating freeze-dried organ products into their wellness routines.

This study is pioneering in its focus on real-world outcomes and the application of scientific rigor to the examination of natural supplementation effects. While individual results may vary, the goal is to offer each participant a tailored understanding of how Whole Package could influence their reproductive health and virility. This could potentially shift the paradigm in male health supplementation, steering away from generic claims towards an evidence-based appreciation of the impact of organ-derived supplements on long-term well-being and performance. Through this research, investigators aspire to equip men with the knowledge to make informed decisions about their health and wellness strategies, ultimately redefining the landscape of male health supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-10-17 (Estimated); Study Completion 2026-10-17 (Estimated)

PRIMARY OUTCOMES:
Men's Health Blood Test | Change from baseline (Day 1-5) in blood test parameters at 11-13 weeks after the start of the intervention
  Efforia, in collaboration with Tasso, introduces the "Comprehensive Men's Health Test," covering Total and Free Testosterone, Albumin, SHBG, PSA, DHEA-S, and Estradiol. Our advanced, shoulder-worn device collects a small blood sample easily and without needles. A bit pricier, yet much less daunting than standard methods, it's perfect for the needle-shy. Simply return it in the included pre-paid envelope for detailed lab analysis. Convenient, eff
AGING MALE SYMPTOMS SCALE (AMS) | Change from baseline (Day 1-5) in AMS score at 11-13 weeks after the start of the intervention
  The Aging Male Symptoms Scale (AMS) is designed to assess various symptoms that may affect aging males, contributing vital information for healthcare providers in managing age-related conditions. This tool is particularly valuable as it encompasses a wide range of physical, emotional, and sexual health issues, enabling targeted interventions. By quantifying the severity of symptoms from "none" to "extreme," the AMS helps in monitoring the progression or improvement of symptoms over time. This structured approach aids in the clinical evaluation and can guide treatment decisions effectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=41342